CLINICAL TRIAL: NCT04984226
Title: Randomized Cross-over Trial of Sodium Bicarbonate on Muscle Mitochondrial Energetics and Physical Endurance in Chronic Kidney Disease and Metabolic Acidosis
Brief Title: Sodium Bicarbonate and Mitochondrial Energetics in Persons With CKD
Acronym: Senergy-CKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Baback Roshanravan, Associate Professor, Nephrology, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1343905; 5R01DK129793 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases; Metabolic Acidosis; Fatigue; Physical Endurance; Insulin Resistance; Mitochondrial Energetics; Diabetes
Keywords: Metabolic acidosis; Chronic kidney disease; Insulin resistance
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis; Fatigue; Insulin Resistance; Diabetes Mellitus | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate 16 weeks (Experimental): Sodium bicarbonate will be dosed at 0.8meq per kilogram of ideal body weight daily (1meq is approximately 84mg). We will use the Devine formula to determine ideal body weight. Investigational Drug Services at both UC Davis and Vanderbilt will compound the sodium bicarbonate. Sodium bicarbonate 650 mg tablets will be over-encapsulated and matching placebo capsules will be prepared. Participants will be limited to a maximum of 9 capsules daily (maximum dose = 5850mg of sodium bicarbonate). Capsules will be dispensed to patients in two separate 8-week allotments. The dose will be rounded to the nearest whole capsule and depending on participant preference may be divided into portions taken twice or thrice daily. Given the high probability of interruption in sodium bicarbonate supply and availability, we may need to change brands of sodium bicarbonate intermittently.
  Interventions: Drug: Sodium bicarbonate
- placebo 16 weeks (Placebo Comparator): Microcrystalline cellulose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate will be dosed at 0.8meq per kilogram of ideal body weight daily (1meq is approximately 84mg). We will use the Devine formula to determine ideal body weight. Investigational Drug Services at both UC Davis and Vanderbilt will compound the sodium bicarbonate. Sodium bicarbonate 650 mg tablets will be over-encapsulated and matching placebo capsules will be prepared. Participants will be limited to a maximum of 9 capsules daily (maximum dose = 5850mg of sodium bicarbonate). Capsules will be dispensed to patients in two separate 8-week allotments. The dose will be rounded to the nearest whole capsule and depending on participant preference may be divided into portions taken twice or thrice daily. Given the high probability of interruption in sodium bicarbonate supply and availability, we may need to change brands of sodium bicarbonate intermittently.
  Arms: Sodium bicarbonate 16 weeks
Drug: placebo — The placebo and filler for for sodium bicarbonate capsules will be comprised of microcrystalline cellulose. Capsule appearance for control and sodium bicarbonate will be the same.
  Arms: placebo 16 weeks

SUMMARY:
Skeletal muscle metabolic health is critical for mobility and an underrecognized target of metabolic acidosis in chronic kidney disease. Impaired muscle mitochondrial metabolism underlies poor physical endurance increasing the risk of mobility disability. The proposed project will use precise in vivo tools to study the pathophysiology of poor physical endurance in a clinical trial treating metabolic acidosis among persons living with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is highly prevalent affecting 14% of the U.S. population leading to substantial morbidity and reduced quality of life. Older adults with CKD identify maintenance of functional independence as their top priority. Skeletal muscle health is critical for mobility and an underrecognized target of metabolic acidosis (MA) and protein energy wasting in CKD. Skeletal muscle endurance provides a window into muscle metabolic health and muscle quality. Muscle mitochondrial metabolism is central to muscle and walking endurance providing energy from carbohydrates and fats to power repeated muscle contraction. Investigators showed metabolic acidosis and muscle adiposity as the major determinants of muscle mitochondrial function.

Metabolic acidosis (MA) is long believed to be the main mechanism leading to skeletal muscle wasting and peripheral insulin resistance in CKD. Skeletal muscle mitochondrial metabolism is considered a principal determinant of peripheral insulin sensitivity and muscle quality, but little is known of the impact of MA on muscle mitochondrial function. Muscle mitochondrial dysfunction leads to defective lipid metabolism augmenting adiposity and lipotoxic intermediates resulting in insulin resistance, low endurance, and muscle atrophy. Using in vivo 31Phosphorus Magnetic Resonance Spectroscopy (31P MRS) investigators showed that the presence and severity of CKD is strongly associated with impaired muscle mitochondrial capacity to generate ATP translating into poor walking endurance. Investigators also showed MA and muscle adiposity are the major determinants of muscle mitochondrial function. Despite the importance of mitochondrial function to muscle health, it is unknown if treatment of MA benefits muscle mitochondrial function, adiposity or endurance in CKD.

The proposed project will use precise, in vivo 31P MRS and gold-standard testing of peripheral insulin sensitivity by hyperinsulinemic euglycemic clamp to probe the pathophysiology of MA and low endurance in a clinical trial of alkali therapy in CKD and MA. We will compare sodium bicarbonate to placebo in a multicenter randomized, cross-over trial design in 80 persons with moderate-severe CKD and MA. First, the efficacy of 4-months of alkali therapy will be tested comparing sodium bicarbonate versus placebo on muscle metabolic health in a randomized crossover trial in MA. Second, we will test the efficacy of 4-months of alkali therapy comparing sodium bicarbonate versus placebo on improving physical endurance in MA. The rationale is that identification of therapeutic targets for low physical endurance will inform the development of pharmacologic interventions. Long term, it is expected that strategies treating MA will improve exercise tolerance enabling effective engagement in lifestyle interventions improving quality of life in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe CKD determined by eGFR <50ml/min per 1.73m2 by CKD EPI equation on at least 2 consecutive occasions.
* Metabolic acidosis defined as bicarbonate level<24 on two consecutive occasions. Bicarbonate level of 24 or less allowed if eGFR<=45ml/min per 1.73m2
* Age 21 to 85 years old

Exclusion Criteria:

* Type 1 diabetes
* Poorly controlled diabetes (HgbA1c>10%)
* History of persistent hyperkalemia (K>5.4)
* History of persistent hypokalemia (K<3.3)
* Uncontrolled blood pressure (>170/100)
* Chronic treatment with renal replacement therapy
* History of aortic dissection or severe valvular heart disease
* Exercise induced angina
* Uncontrolled cardiac dysrhythmia
* Oxygen dependent chronic obstructive pulmonary disease (COPD)
* Symptomatic claudication
* End stage liver disease
* Mobility disability defined as inability to walk without human assistance
* Dementia or psychosis
* Patients who cannot consent
* Active use of intraveneous drugs
* Non-english speaking
* History of transplant
* Implants that prohibit MRI measurements or trauma involving metal fragments
* Pacemaker
* Expectation to start dialysis during the course of study.
* Women who are breastfeeding, pregnant, or are wanting to become pregnant
* Any condition which in the judgement of the clinical investigator places the participant at risk from participation in the study.

Exclusion criteria for optional muscle biopsy

* Drugs- anticoagulants or antiplatelets:

  * Anticoagulants, any 1 (coumadin, rivaroxaban, apixaban, dabigatran, edoxaban)
  * Antiplatelets, any 2 (aspirin, cilostazol, clopidogrel, dipyridamole, prasugrel, ticragrelor, ticlopidine, vorapaxar)
* Platelet count <100,000
* International normalized ratio (INR)>1.4

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
muscle mitochondrial oxidative capacity by 31P MRS | 16 weeks
  We will use 31P MRS to evaluate the concentration of phospho-creatine (PCr) and other phosphate-energy carrier molecules in limb muscles. After one minute of basal resting measurements, patients will be asked to perform two knee extensions every second against ankle weights 5-10% of the maximal voluntary contraction. The exercise protocol will last 60-90 seconds (a total of 60 knee extensions) followed by 6 minutes of rest. The intensity of the exercise decreases phosphocreatine (PCr) levels with minimal change in muscle pH. Spectra analysis was performed with AMARES from the jMRUI software package. Spectra are used to calculate the relative concentrations of inorganic phosphate (Pi), PCr, and ATP. PCr recovery will be measured through 6min of rest and fit with a monoexponential equation.
Insulin sensitivity (SI) by insulin clamp | 16 weeks
  Primary endpoint for the hyperinsulinemic euglycemic clamp testing will be insulin sensitivity defined as (glucose disposal rate - concentration of infused glucose)/(insulin concentration at steady state - fasting insulin concentration). Units are mg/min per microunit per milliliter.
total work performed on cycle ergometry VO2 | 16 weeks
  Total work will be obtained by cycle ergometry using standard protocol measuring oxygen uptake starting at 0 watts (W) at 60 rotations per minute (rpm) increasing by 25W every 2 minutes until volitional exhaustion adapting a prior protocol used in CKD patients. The primary measure will be total work completed (Joules).
muscle work efficiency cycle ergometry | 16 weeks
  joules/ml Oxygen(VO2 peak)
Walking endurance by 6-minute walk | 16 weeks
  Meters
FACIT-F Fatigue (PRO) | 16 weeks
  score on FACIT-F questionnaire

SECONDARY OUTCOMES:
Intermuscular fat by MRI | 16 weeks
  Percent intermuscular fat.
30 second sit to stand test | 16 weeks
  number of times patient can get up from sitting position over 30 seconds
PROMIS Fatigue (PRO) | 16 weeks
  score on NIH PROMIS Fatigue questionnaire

OTHER OUTCOMES:
Muscle mitochondrial respiration from in situ high resolution respirometry of muscle biopsy tissue | 16 weeks
  We will determine mitochondrial respiration and oxidative stress under different respiratory states including subsaturating and saturating ADP (state 3), using a combination of complex I (glutamate + malate) and complex II (succinate) substrates, state 4 respiration (proton leak in the absence of ADP and the presence of oligomycin), and fully uncoupled respiration using FCCP. The assay for mtH2O2 production is based on the rate of production of the fluorescent molecule, resorufin, when Amplex Red reacts with H2O2 as described. We a priori select mtH2O2 of reverse electron transport (succinate as substrate in the absence of ADP) as our primary endpoint given the evidence that complex I is the predominant source of mtROS during aerobic exercise. Units are pmol/sec.
Inflammatory cytokines. TNF-alpha and IL-6 | 16 weeks
  Inflammatory cytokines. Units pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Baback Roshanravan, MD, Principal Investigator — UC Davis; Jorge Gamboa, MD PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of California Davis Health, Sacramento, California
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other investigators on request. The requests will include a proposal outlining the research question, specific exposures, outcomes of interest and analytic plan. All requests will be reviewed by the study principal investigators and coinvestigators prior to release of data. All data will be de-identified.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: within 18 months after the conclusion of the study. This data will be available indefinitely